CLINICAL TRIAL: NCT00711490
Title: Pilot Study of the Evaluation of Sirolimus in the Treatment of Diabetic Macular Edema
Brief Title: Sirolimus to Treat Diabetic Macular Edema
Acronym: SDME
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080175; 08-EI-0175
Record Dates: First submitted 2008-07-08; First posted 2008-07-09 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2016-09

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Macular Edema; Diabetic Retinopathy; Rapamycin; Sirolimus; Diabetes
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): The study eye was treated with sirolimus.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — 20 μL (440 μg) of sirolimus were injected at baseline, Month 2, and every 2 months thereafter if re-treatment criteria were satisfied.
  Other Names: Rapamune

SUMMARY:
Objective: Diabetic macular edema (DME) is a frequent manifestation of diabetic retinopathy, a leading cause of blindness in the United States. The only proven treatment for DME is laser photocoagulation. Sirolimus has been shown to inhibit the production, signaling and activity of many growth factors relevant to the development of diabetic retinopathy. Therefore, this study will investigate the safety and efficacy of multiple sirolimus injections in patients with DME.

Study Population: Eligibility criteria include central macular thickening > 260 microns and visual acuity 20/32 or worse in one or both eyes.

Design: Five participants will be enrolled into this open-label pilot study. After receiving a 20 μL (440 μg) subconjunctival injection in the study eye at baseline and Month 2, the participants will be re-evaluated every two months for at least one year for possible additional injections. During follow-up, participants will not undergo re-injection if they show significant clinical improvement or treatment success, defined as no intraretinal fluid or cysts present on optical coherence tomography (OCT) OR 100% reduction in excess retinal thickness over 260 microns on OCT OR no leakage on fluorescein angiography (FA). Beginning at Month 4, participants will be assessed for treatment failure, defined as loss of 15 or more letters of vision compared to baseline at two consecutive visits OR a 50% or greater increase in total retinal thickness as measured by OCT at two consecutive visits. Individual participants deemed treatment failures will continue receiving sirolimus injections, but will be allowed to receive focal laser therapy for any amenable leaking microaneurysms at Month 4. Beginning at Month 6, focal laser therapy will be permitted for both treatment failures and participants who do not meet the criteria of a treatment success. Participants will have the option of continuing treatment until a common termination date of one year.

Outcome Measures: The primary outcome is the change in visual acuity in the study eye at six months compared to baseline. Secondary outcomes include changes in visual acuity in the study eye at one year as compared with baseline, changes in retinal thickness as measured by OCT and changes in fluid leakage in the macula as demonstrated by FA at six months, one year and throughout the study period in the study and fellow eyes. Safety outcomes include number and severity of systemic and ocular toxicities, adverse events and infections, and the number of participants withdrawn from study therapy.

ELIGIBILITY:
Participant-Level Inclusion Criteria

1. Participant is 18 years of age or older.
2. Diagnosis of diabetic mellitus (type 1 or type 2).

   Any one of the following will be considered to be sufficient evidence that diabetes is present:
   1. Current regular use of insulin for the treatment of diabetes.
   2. Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes.
   3. Documented diabetes by American Diabetes Association (ADA) and/or World Health Organization (WHO) criteria.
3. Documented hemoglobin A1C 12% or less within one month of baseline.
4. Able and willing to provide informed consent.
5. Both female participants of childbearing potential and male participants able to father a child must agree to practice two* forms of adequate birth control throughout the course of the study and for three months following the completion of the study treatment. Acceptable methods of birth control include hormonal contraception (birth control pills, injected hormones or vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom and spermicide) or surgical sterilization (hysterectomy, tubal ligation or vasectomy).

   *Participants with a hysterectomy or vasectomy (or who have a partner with a hysterectomy or vasectomy) are exempt from using two methods of contraception. However, female participants with a tubal ligation (or male participants who have a female partner with a tubal ligation) are not exempt, and are required to practice another acceptable method of birth control.
6. Female participants of childbearing potential must be willing to undergo pregnancy testing for the duration of the study.
7. At least one eye meets the study eye criteria listed in Section 4.2.

Participant-Level Exclusion Criteria

1. History of chronic renal failure requiring dialysis or kidney transplant.
2. Positive serum or urine pregnancy test or currently lactating for women of childbearing potential.
3. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).
4. Participation in an investigational trial within 30 days of study entry that involved treatment with any drug that has not received regulatory approval at the time of study entry.
5. History of cancer (other than a non-melanoma skin cancer) diagnosed within the past five years that could be worsened by immunosuppression.*

   *The risk of immunosuppression must be determined by an oncology consultation prior to enrollment.
6. Laboratory values outside normal limits and considered clinically significant by the investigator.
7. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110).
8. History of intravitreal anti-VEGF therapy or subtenon/intravitreal steroids in either eye within three months prior to study entry.
9. History of treatment with systemic anti-VEGF agents or steroids within one year prior to study entry.
10. Participant is currently taking one of the following drugs: amprenavir, atazanavir, clarithromycin, darunavir, delavirdine, erythromycin, fluconazole (at doses of 200mg or greater), fluvoxamine, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, quinupristin, ritonavir, saquinavir, telithromycin, troleandomycin, verapamil or voriconazole.

Study Eye Inclusion Criteria

1. Best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity score of ≤ 74 letters (i.e., 20/32 or worse).
2. Definite retinal thickening due to diabetic macular edema based on clinical exam involving the center of the macula that is not refractory to further therapy as based on the investigator's clinical judgment.
3. Retinal thickness on baseline OCT measurement > 260 microns in the central subfield.
4. Media clarity, pupillary dilation and patient cooperation sufficient for adequate fundus photographs.

Study Eye Exclusion Criteria

1. Macular edema is considered to be due to a cause other than diabetic macular edema.
2. An ocular condition is present such that, in the opinion of the investigator, visual acuity would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentary changes, dense subfoveal hard exudates, nonretinal condition, etc.).
3. An ocular condition is present (other than diabetic retinopathy) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, Irvine-Gass Syndrome, etc.).
4. Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by three lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).
5. History of focal/grid macular photocoagulation within 12 weeks (three months) prior to study entry.
6. History of panretinal scatter photocoagulation (PRP) within four months prior to study entry.
7. Anticipated need for PRP in the four months following study entry.
8. History of prior pars plana vitrectomy.
9. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior six months or anticipated within the next six months following study entry.
10. History of (Yttrium Aluminium Garnet) YAG laser capsulotomy performed within two months prior to study entry.
11. Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant blepharitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Meyerle, MD, Principal Investigator — National Eye Institute/ National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kempen JH, O'Colmain BJ, Leske MC, Haffner SM, Klein R, Moss SE, Taylor HR, Hamman RF; Eye Diseases Prevalence Research Group. The prevalence of diabetic retinopathy among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):552-63. doi: 10.1001/archopht.122.4.552. PMID 15078674
- [Background] Klein R, Klein BE, Moss SE, Davis MD, DeMets DL. The Wisconsin epidemiologic study of diabetic retinopathy. IV. Diabetic macular edema. Ophthalmology. 1984 Dec;91(12):1464-74. doi: 10.1016/s0161-6420(84)34102-1. PMID 6521986
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Result] Krishnadev N, Forooghian F, Cukras C, Wong W, Saligan L, Chew EY, Nussenblatt R, Ferris F 3rd, Meyerle C. Subconjunctival sirolimus in the treatment of diabetic macular edema. Graefes Arch Clin Exp Ophthalmol. 2011 Nov;249(11):1627-33. doi: 10.1007/s00417-011-1694-9. Epub 2011 May 13. PMID 21567211

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus: This is a single-arm study with all participants receiving a minimum of two 20 μL (440 μg) sirolimus injections: one injection at baseline and one injection at Month 2. Patients for whom re-treatment criteria were satisfied received additional injections every 2 months thereafter.
Period: Overall Study
Arm/Group | Sirolimus
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Acuity From Baseline to 6 Months
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. This acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters the Snellen measurement is 20/20.
Time Frame: 6 months
Measure: Median (Full Range); unit: ETDRS letters
Groups:
- Study Eye: The study eye was treated with sirolimus.
- Fellow Eye: The fellow eye was not treated with sirolimus.
Arm/Group | Study Eye | Fellow Eye
Number analyzed (Participants) | 5 | 5
ETDRS letters | 7 [-7 to 13] | 0 [-4 to 2]

2. Secondary Outcome: Change in Visual Acuity From Baseline to 12 Months
Description: as for outcome 1
Time Frame: 12 months
Measure: Median (Full Range); unit: ETDRS letters
Arm/Group | Study Eye | Fellow Eye
Number analyzed (Participants) | 5 | 5
ETDRS letters | 1 [-8 to 13] | -1 [-3 to 1]

3. Secondary Outcome: Change in Retinal Thickness From Baseline to 6 Months, as Measured by Optical Coherence Tomography (OCT)
Description: Retinal thickness was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue.
Time Frame: 6 months
Measure: Median (Full Range); unit: μm
Arm/Group | Study Eye | Fellow Eye
Number analyzed (Participants) | 5 | 5
μm | -37 [-163 to 74] | -10 [-63 to 0]

4. Secondary Outcome: Change in Retinal Thickness From Baseline to 12 Months, as Measured by Optical Coherence Tomography (OCT)
Description: as for outcome 3
Time Frame: 12 months
Measure: Median (Full Range); unit: μm
Arm/Group | Study Eye | Fellow Eye
Number analyzed (Participants) | 5 | 5
μm | -55 [-321 to 144] | -51 [-152 to -7]

5. Secondary Outcome: Change in Fluid Leakage in the Macula of the Study Eye From Baseline to 6 Months, as Measured on Fluorescein Angiography (FA)
Time Frame: 6 months
Population: Due to lack of effect in other outcome measures, at investigator's discretion, data for this outcome measure was neither collected nor analyzed. As such, zero participants have data for this outcome.
Arm/Group | Study Eye
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Fluid Leakage in the Macula of the Study Eye From Baseline to 12 Months, as Measured on Fluorescein Angiography (FA)
Time Frame: 12 months
Population: as for outcome 5
Arm/Group | Sirolimus
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Duration of study
Arm/Group | Sirolimus
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=5)
Blood urea increased (Investigations) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4)
White blood cell count decreased (Investigations) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Oedema peripheral (General disorders) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Blood cholesterol increased (Investigations) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Blood glucose increased (Investigations) | 2 (2)
Blood uric acid increased (Investigations) | 2 (2)
Glycosylated haemoglobin increased (Investigations) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Red cell distribution width increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (4)
Blood trigylcerides increased (Investigations) | 2 (2)
Conjunctival hyperaemia (Eye disorders) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Red blood cell count decreased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (2)
Blood pressure increased (Investigations) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Blood chloride increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes